CLINICAL TRIAL: NCT03307226
Title: Suubi4Her: A Combination Intervention Addressing HIV Risk Behaviors Among Older Adolescent Girls Transitioning Into Adulthood in Uganda
Brief Title: Suubi4Her: Combination Intervention for Adolescent Girls Transitioning Into Adulthood in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201703102; 1R01MH113486-01 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS
Keywords: Suubi; Adolescent Girls; Poverty; Economic Empowement Interventions; Adherence to HIV antiretroviral therapy; HIV/AIDS-impacted girls; Uganda; Cost-effectiveness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Youth Development Accounts (YDA) (Experimental): Youth Development Accounts (YDA)
  * Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development
  * Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs) Behavioral: Youth Development Accounts (YDA)
  Interventions: Behavioral: Youth Development Accounts (YDA)
- YDA + Multiple Family Groups (MFG) (Experimental): YDA + Multiple Family Groups (MFG)
  * Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development
  * Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs)
  * Multiple Family Groups sessions focused on strengthening family relationships and mental health
  Interventions: Behavioral: YDA + Multiple Family Groups (MFG)
- Usual Care (No Intervention): Usual Care consisting of curricula delivered at secondary schools in Uganda including Life Planning Skills, and Adolescent Sexual Reproductive Health

INTERVENTIONS:
Behavioral: Youth Development Accounts (YDA) — Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs) Behavioral: Youth Development Accounts (YDA)
  Arms: Youth Development Accounts (YDA)
Behavioral: YDA + Multiple Family Groups (MFG) — Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development 12 Financial Management workshops on asset-building, saving and investing in Income Generating Activities (IGAs) 18 Multiple Family Groups sessions focused on strengthening family relationships and mental health
  Arms: YDA + Multiple Family Groups (MFG)

SUMMARY:
This study examines the impact and cost associated with Suubi4Her, an innovative combination intervention that aims to prevent HIV risk behaviors among 15-17 year-old girls living in communities heavily affected by poverty and HIV/AIDS in Uganda. Participants will be randomly assigned at the school level into one of three study conditions: 1) Savings (Youth Development Accounts - YDA) - with a 1:1 incentive match rate - for education and microenterprise development; 2) Savings (YDA) + Multiple Family Groups intervention; 3) Control condition receiving standard health and sex education provided in schools. The intervention will last for 24 months. Assessments will be conducted at baseline, 12, 24 and 36 months. Assessments will include biologically confirmed STIs, proportion of HIV infections during the study period, and for HIV+ participants markers for ART adherence. The study aims to examine the impact of the Suubi4Her intervention on behavioral health functioning, and protecting adolescent girls against known HIV risk factors. The study will also examine the cost-effectiveness of each intervention condition.

DETAILED DESCRIPTION:
Aligned with the NIH priority of addressing disparities in new HIV infections and the UNAIDS call for implementing combination HIV prevention approaches, the proposed study will examine the impact and cost associated with Suubi4Her, an innovative combination intervention that aims to prevent HIV risk behaviors among 14-17 year-old girls living in communities heavily affected by poverty and HIV/AIDS in Uganda. In sub-Saharan Africa (SSA), family financial stress can compromise the support available to adolescents, with girls living in poverty exhibiting higher rates of risky sexual behavior increasing their vulnerability in acquiring HIV and other STIs. At the same time, internalizing mental health disorders such as depression and low self-esteem disproportionately affect girls and may be contributing to HIV risk behavior. Against that backdrop, support over and above health and sex education is needed to help adolescent girls in SSA successfully transition into young adulthood. The proposed study is informed by two previously tested interventions - asset-based matched savings accounts (YDA) and family strengthening through Multiple Family Groups (MFG) which have successfully been implemented with younger primary school-going adolescents. Suubi4Her will test the theory that youth cognitive and behavioral change is influenced by economic stability while examining if enhanced intra-familial support and communication are needed to maintain positive behavioral health functioning and reinforce engagement in protective health behaviors. Nested within 47 secondary schools across four districts of Uganda heavily impacted by HIV/AIDS, 1260 older girls (ages 14-17 at enrollment) will be randomly assigned (at school level) to one of three study conditions: 1) Savings (Youth Development Accounts - YDA)- with a 1:1 incentive match rate - for education and microenterprise development; 2) Savings (YDA) + MFG intervention; 3) Control condition receiving standard health and sex education provided in schools. The intervention will be provided for 24 months. Assessments at baseline,12, 24, and 36-months will include biomedical data to measure our primary sexual-risk outcome:1) proportion of girls' biologically confirmed STIs (Gonorrhea, Trichomonas and Chlamydia); and secondary outcomes: 2) the proportion of new HIV infections during the study period, and 3) for HIV+ girls, viral load and CD4 as markers of ART adherence. The study aims are to: 1) Examine whether the Suubi4Her intervention is effective in protecting adolescent girls against known HIV risk factors (including economically-motivated sex and intimate partner violence). 2) Elucidate the effects of the Suubi4Her intervention on behavioral health functioning (i.e., depression, self-efficacy and hopelessness) and examine the effects of these variables as potential mechanisms of change, mediating the relationship between each intervention and HIV risk reduction. 3) Evaluate the cost-effectiveness of each intervention condition. The study will also use the Child Depression Index and Beck Hopelessness Scale to examine the efficacy of interventions in improving mental health in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

(1) female; (2) enrolled in first year of secondary school in Rakai, Masaka, Lwengo or Kalungu districts; (3) age 14-17 years; (4) living within a family (broadly defined and not an institution or orphanage, as those in institutions have different familial needs)

Exclusion Criteria:

(5) they have a cognitive or severe psychiatric impairment that would prevent comprehension of study procedures as assessed during the Informed Consent process or; (6) they are unwilling or unable to commit to completing the study.

We will not exclude girls because of their HIV, STI and/or pregnancy status. Analysis will be adjusted to account for these baseline factors. Girls testing positive for HIV, STI or pregnancy will be referred for care and support.

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants must be female.
Enrollment: 1260 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Ssewamala, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- International Center for Child Health and Development, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per CFR Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Columbia University School of Social Work Office of Sponsored Projects' data sharing agreement.

REFERENCES:
- [Derived] Ssewamala FM, Tozan Y, Brathwaite R, Kiyingi J, Namatovu P, Bahar OS, Nabunya P, Nartey PB, Neilands TB. Cost-Effectiveness of an Economic Empowerment and Family Intervention on Mental Health Among School-Going Adolescent Girls in Uganda, 2017-2022. Am J Public Health. 2025 Sep;115(9):1408-1416. doi: 10.2105/AJPH.2025.308135. Epub 2025 Jun 26. PMID 40570278
- [Derived] Karimli L, Nabunya P, Ssewamala FM, Dvalishvili D. Combining Asset Accumulation and Multifamily Group Intervention to Improve Mental Health for Adolescent Girls: A Cluster-Randomized Trial in Uganda. J Adolesc Health. 2024 Jan;74(1):78-88. doi: 10.1016/j.jadohealth.2023.08.012. Epub 2023 Sep 16. PMID 37715767
- [Derived] Filiatreau LM, Tutlam N, Brathwaite R, Byansi W, Namuwonge F, Mwebembezi A, Sensoy-Bahar O, Nabunya P, Neilands TB, Cavazos-Rehg P, McKay M, Ssewamala FM. Effects of a Combination Economic Empowerment and Family Strengthening Intervention on Psychosocial Well-being Among Ugandan Adolescent Girls and Young Women: Analysis of a Cluster Randomized Controlled Trial (Suubi4Her). J Adolesc Health. 2023 May;72(5S):S33-S40. doi: 10.1016/j.jadohealth.2022.11.250. PMID 37062582
- [Derived] Byansi W, Ssewamala FM, Neilands TB, Mwebembezi A, Nakigozi G. Patterns of and Factors Associated With Mental Health Service Utilization Among School-Going Adolescent Girls in Southwestern Uganda: A Latent Class Analysis. J Adolesc Health. 2023 May;72(5S):S24-S32. doi: 10.1016/j.jadohealth.2022.09.037. PMID 37062580
- [Derived] Sensoy Bahar O, Nabunya P, Namuwonge F, Samtani S, Ssentumbwe V, Namuli F, Magorokosho N, Ssewamala FM. "It gives you a road map of what to do to solve your problems": acceptability of a combination HIV prevention intervention among adolescent girls in Uganda. BMC Public Health. 2023 Feb 6;23(1):249. doi: 10.1186/s12889-023-15083-2. PMID 36747149
- [Derived] Ssewamala FM, Brathwaite R, Neilands TB. Economic Empowerment, HIV Risk Behavior, and Mental Health Among School-Going Adolescent Girls in Uganda: Longitudinal Cluster-Randomized Controlled Trial, 2017-2022. Am J Public Health. 2023 Mar;113(3):306-315. doi: 10.2105/AJPH.2022.307169. Epub 2023 Jan 5. PMID 36603167
- [Derived] Byansi W, Ssewamala FM, Neilands TB, Sensoy Bahar O, Nabunya P, Namuwonge F, McKay MM. The Short-Term Impact of a Combination Intervention on Depressive Symptoms Among School-Going Adolescent Girls in Southwestern Uganda: The Suubi4Her Cluster Randomized Trial. J Adolesc Health. 2022 Sep;71(3):301-307. doi: 10.1016/j.jadohealth.2022.04.008. Epub 2022 Jun 1. PMID 35660128
- [Derived] Nabunya P, Damulira C, Byansi W, Muwanga J, Bahar OS, Namuwonge F, Ighofose E, Brathwaite R, Tumwesige W, Ssewamala FM. Prevalence and correlates of depressive symptoms among high school adolescent girls in southern Uganda. BMC Public Health. 2020 Nov 25;20(1):1792. doi: 10.1186/s12889-020-09937-2. PMID 33238965
- [Derived] Ssewamala FM, Bermudez LG, Neilands TB, Mellins CA, McKay MM, Garfinkel I, Sensoy Bahar O, Nakigozi G, Mukasa M, Stark L, Damulira C, Nattabi J, Kivumbi A. Suubi4Her: a study protocol to examine the impact and cost associated with a combination intervention to prevent HIV risk behavior and improve mental health functioning among adolescent girls in Uganda. BMC Public Health. 2018 Jun 5;18(1):693. doi: 10.1186/s12889-018-5604-5. PMID 29871619

RESULTS

PARTICIPANT FLOW:
Groups:
- Youth Development Accounts (YDA): Youth Development Accounts (YDA)
  * Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development
  * Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs) Behavioral: Youth Development Accounts (YDA)
  Youth Development Accounts (YDA): Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs) Behavioral: Youth Development Accounts (YDA)
- YDA + Multiple Family Groups (MFG): YDA + Multiple Family Groups (MFG)
  * Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development
  * Financial workshops on asset-building, saving and investing in Income Generating Activities (IGAs)
  * Multiple Family Groups sessions focused on strengthening family relationships and mental health
  YDA + Multiple Family Groups (MFG): Youth Development Accounts (YDA) with 1:1 incentive match rate to be used for education and microenterprise development 12 Financial Management workshops on asset-building, saving and investing in Income Generating Activities (IGAs) 18 Multiple Family Groups sessions focused on strengthening family relationships and mental health
Period: Overall Study
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Started | 471 | 381 | 408
Completed | 441 | 344 | 380
Not Completed | 30 | 37 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care | Total
Number analyzed (Participants) | 471 | 381 | 408 | 1260
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (0.8) | 15.4 (0.9) | 15.2 (0.9) | 15.4 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 471 | 381 | 408 | 1260
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 471 | 381 | 408 | 1260
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 471 | 381 | 408 | 1260

OUTCOME MEASURES:

1. Primary Outcome: Proportion With STIs From Baseline to Follow-up Assessments
Description: Proportion of girls biologically confirmed STIs (Gonorrhea, Tirchomonas, and Chlamydia) or positive pregnancy test at each assessment time point (Baseline, 12-, 24-, and 36-month follow-up)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Number analyzed (Participants) | 471 | 381 | 408
Participants
  Number of girls biologically confirmed positive for STIs or positive pregnancy test at Baseline | 43 | 20 | 29
  Number of girls biologically confirmed negative for STIs or positive pregnancy test at baseline | 428 | 361 | 379

2. Primary Outcome: Proportion With STIs From Baseline to Follow-up Assessments
Description: Proportion of girls biologically confirmed STIs (Gonorrhea, Trichomonas, and Chlamydia) or positive pregnancy test at each assessment time point (Baseline, 12-, 24-, and 36-month follow-up)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Number analyzed (Participants) | 457 | 366 | 396
Participants
  Proportion of girls biologically confirmed positive for STIs or positive pregnancy test at 12 months | 22 | 22 | 15
  Proportion of girls biologically confirmed negative for STIs or positive pregnancy test at 12 months | 435 | 344 | 381

3. Secondary Outcome: Proportion Positive for HIV Infections at Each Assessment Time Point (Baseline, 12-, 24-follow-up)
Description: Proportion positive for HIV at baseline
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Number analyzed (Participants) | 471 | 381 | 408
Participants
  Number positive for HIV | 3 | 1 | 4
  Number negative for HIV | 468 | 380 | 404

4. Secondary Outcome: Change in Adherence to HIV Treatment From Baseline to Follow-up Assessments
Description: For HIV+ participants, adherence to HIV treatment regimen outcomes as measured through viral load and CD4 counts
Time Frame: baseline
Population: Viral load and CD4 data were not collected and hence the data cannot be reported.
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Cost-Effectiveness Analyses
Description: Cost-effectiveness analyses measuring the cost of achieving an agreed upon benefit, such as an additional year of schooling, employment, or a reduction in a disease. Costs will be measured on a per person basis. The costs of the intervention will include all program costs. Research costs will not be included.
Time Frame: Every year for five years
Reporting Status: Not Posted, anticipated posting 2025-02

6. Secondary Outcome: Proportion Positive for HIV Infections at Each Assessment Time Point (Baseline, 12-, 24-follow-up)
Description: Proportion Positive for HIV Infections at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
Number analyzed (Participants) | 457 | 366 | 396
Participants
  Number positive for HIV | 4 | 2 | 4
  Number negative for HIV | 453 | 364 | 392

ADVERSE EVENTS:
Time Frame: baseline, 12 months, 24 months
Arm/Group | Youth Development Accounts (YDA) | YDA + Multiple Family Groups (MFG) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/471 | 1/381 | 0/408
Serious Adverse Events (participants affected / at risk) | 0/471 | 0/381 | 0/408
Other Adverse Events (participants affected / at risk) | 0/471 | 0/381 | 0/408

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03307226/Prot_SAP_000.pdf